CLINICAL TRIAL: NCT03574922
Title: The Effects of Core Stabilization Exercises in Addition to Balance Exercises in Adult Hemophilia Patients on Balance, Quality of Life, Lower Limb Muscle Strength and Functional Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sercan ONAL, MSc., PT., Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA-17161
Record Dates: First submitted 2018-05-02; First posted 2018-07-02 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-05

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Balance Exercises (Active Comparator): Balance Exercises
  Interventions: Other: Balance exercises; Other: Core Stabilization exercises
- Core Stabilization Exercises (Active Comparator): Balance and core stabilization exercises
  Interventions: Other: Balance exercises; Other: Core Stabilization exercises
- Control (No Intervention): Assessments only

INTERVENTIONS:
Other: Balance exercises — Balance Exercises
  Arms: Balance Exercises; Core Stabilization Exercises
Other: Core Stabilization exercises — Core Stabilization exercises
  Arms: Balance Exercises; Core Stabilization Exercises

SUMMARY:
The aim of this study is to investigate the effects of core stabilization exercises in addition to balance exercises on balance, quality of life, lower extremity muscle strength and functional level in adult hemophilic patients.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of core stabilization exercises in addition to balance exercises on balance, quality of life, lower extremity muscle strength and functional level in adult hemophilic patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia Patients

Exclusion Criteria:

* Acute Bleeding

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Balance Tests | 8 Weeks
  Functional Reach Test

SECONDARY OUTCOMES:
Functionality Tests | 8 Weeks
  Timed up and go

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Can, Principal Investigator — Hacettepe University
Locations (1):
- Sercan Aykar, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided